CLINICAL TRIAL: NCT02206009
Title: PriMatrix Dermal Repair Scaffold Utilization Intraorally
Brief Title: Use of a Collagen Membrane for Soft Tissue Grafting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lauren M. F. Syrowik (Other)
Responsible Party: Sponsor-Investigator, Lauren M. F. Syrowik, DDS, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-000767
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Localized Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Collagen membrane (Experimental): First, the recipient site is prepared, and the collagen membrane hydrated. The collagen membrane is sutured firmly against the prepared vascular bed with a long-lasting suture material. The subject is requested to minimize the amount of manipulation to the area to maintain graft stability.
  Interventions: Device: Collagen Membrane

INTERVENTIONS:
Device: Collagen Membrane — First, the recipient site is prepared, and the collagen membrane hydrated. The collagen membrane is sutured firmly against the prepared vascular bed with a long-lasting suture material. The subject is requested to minimize the amount of manipulation to the area to maintain graft stability.
  Other Names: PriMatrix

SUMMARY:
Is PriMatrix wound dressing capable of regenerating gum tissue inside the mouth?

DETAILED DESCRIPTION:
PriMatrix is an acellular fetal bovine dermal matrix that has a wide array of FDA approved uses. These uses include partial- and full-thickness wounds, pressure, diabetic, and venous ulcers, surgical wounds, trauma wounds, tunneled wounds, and draining wounds. It is a sheet-like matrix made up primarily of type I and type III collagen. An increased proportion of type III collagen appears to play a key role in healing and regeneration.

The use of extracellular dermal matrices is a relatively young field, and the exact mechanism by which PriMatrix promotes skin regeneration is still unknown. Despite this, PriMatrix has demonstrated differences in manufacturing and molecular composition that make it conducive to the harsh environments in which it has already been tested. Intraorally, where there is a rich vascular bed, this material holds exceeding promise.

Utilizing this vascularity, autogenous free gingival grafts from the palate have already had their efficacy proven as a method of augmenting the keratinized tissue.The need to increase the keratinized tissue is based upon the postulation that less mobile, keratinized epithelium is more resilient than the non-keratinized oral mucosa. This is especially important in areas where recession and attachment loss has already occurred. Without having keratinized gingiva apical to the recession area, it has been suggested that there is a greater risk for more attachment loss to occur, thus reducing the support for the tooth. In addition, autogenous free gingival grafts have demonstrated the phenomenon of "creeping attachment" where a portion of the recession actually becomes covered as a result of grafting.

While autogenous grafting is the gold standard in soft tissue augmentation, the amount of tissue that can be taken from the palate is limited, making it difficult to treat patients with generalized recession. Furthermore, a secondary surgical site increases the morbidity associated with the procedure. The hypothesis of this study is that PriMatrix will be able to provide similar results to an autogenous free gingival graft.

ELIGIBILITY:
Inclusion Criteria:

* Must have one to three consecutive teeth with recession and less than 1 mm of keratinized gingiva

Exclusion Criteria:

* Asthma
* Pregnancy
* Uncontrolled diabetes
* Use of continuous positive airway pressure (CPAP) machine for sleep apnea
* Oral appliances (removable partial dentures, braces, mandibular advancement, bruxism splints, etc.)
* Tobacco use
* Immunocompromised individual

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in depth of keratinized tissue | baseline, approximately 6 months after the procedure
  The amount of gingival augmentation will be assessed by the depth of keratinized tissue, measured in millimeters. Change in the amount of keratinized tissue in the areas of interest from baseline to 6 months will be tested to see if they are statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Assad, DDS, Study Director — Mayo Clinic; Lauren MF Syrowik, DDS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States